CLINICAL TRIAL: NCT03993119
Title: Non-Interventional, Cross-sectional Study to Describe NOACs Management in Elderly Patients With Non-valvular Atrial Fibrillation (NVAF) in Spain.
Brief Title: This Study Observes the Usage of Non-vitamin K Antagonist Oral Anticoagulants (NOACs) in Elderly Patients With a Heart Rhythm Disorder in Spain
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0297
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with NVAF
  Interventions: Drug: Non-vitamin K antagonist oral anticoagulant

INTERVENTIONS:
Drug: Non-vitamin K antagonist oral anticoagulant — Non-vitamin K antagonist oral anticoagulant

SUMMARY:
This is an observational, multicenter and cross-sectional study in Non-valvular atrial fibrillation (NVAF) elderly patients currently on Non-vitamin K antagonist oral anticoagulant (NOAC) treatment for their stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients are willing and provide written informed consent prior to participate in this study
* Patients ≥ 75 years-old at the time of the study visit.
* Patients with a diagnosis of non-valvular atrial fibrillation (NVAF).
* Patients who are being treated with NOAC treatment according to the indication approved in the Summary of Product Characteristics (SmPC).
* Patients who have started the NOAC treatment at least 3 months prior to the study visit.

Exclusion Criteria:

Patients will be excluded from participating in this study if the following criterion is met:

* Current participation in any clinical trial of a drug or device.
* Patients who have any contraindication for NOAC treatment, according to the SmPC.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Approximately 500 elderly patients with NVAF currently on NOAC treatment are planned to be included in the study. To minimize selection bias at the patient level, consecutive patients from each site who meet entry criteria will be enrolled. It is planned to have a 9-month recruitment period from first site initiated, or until the sample size is achieved.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia canals, (+34) 93 404 58 77, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (45):
- Spain (45):
  - H. Fundación Alcorcón, Alcorcón, Madrid
  - Consulta Privada, Almería
  - H. Dr. José Molina Orosa, Arrecife, Las Palmas
  - Centro Médico San Juan de Dios, Barakaldo, Bizkaia
  - H. Sagrat Cor, Barcelona
  - H. Vall d'Hebron, Barcelona
  - H. Sant Pau, Barcelona
  - H. Vithas Internacional Xanit, Benalmádena, Málaga
  - Ambulatorio Txurdinaga, Bilbao
  - H. San Juan de Dios de Bormujos, Bormujos, Sevilla
  - H. Provincial de Castellón, Castellon
  - H. San Pedro Alcántara, Cáceres
  - Consulta privada Dr. Ruiz, Córdoba
  - H. Arquitecto Marcide, Ferrol, A Coruña
  - H. de Jaen, Jaén
  - H. U. de León, León
  - H. Arnau de Vilanova, Lleida
  - H. Lucus Augusti, Lugo
  - H. La Princesa, Madrid
  - Sanitas La Zarzuela, Madrid
  - H. Central de la Defensa Gómez, Madrid
  - H. Puerta de Hierro, Majadahonda, Madrid
  - H. de Mataró, Mataró, Barcelona
  - Consulta Privada, Málaga
  - H. de Mendaro, Mendaro, Guipúzcoa
  - H. Morales Meseguer, Murcia
  - H. Virgen de la Arrixaca, Murcia
  - Consulta privada Merelles Otero, Ourense
  - Consulta Privada, Ourense
  - H. Río Carrión, Palencia
  - H. Son Llatzer, Palma de Mallorca
  - H. de Navarra, Pamplona
  - H. Comarcal de la Vega Baja, San Bartolomé, Alicante
  - H. Moises Broggi, Sant Joan Despí, Barcelona
  - H. Marqués de Valdecilla, Santander
  - H. Álvarez-Buylla, Santullano, Asturias
  - H. Virgen de la Macarena, Seville
  - H. Virgen del Valle, Toledo
  - H. de Torrejón, Torrejón de Ardoz, Madrid
  - Consulta Privada, Valencia
  - H. General de Valencia, Valencia
  - Hospital La Fe, Valencia
  - H. Virgen de la Concha, Zamora
  - H. Clínico Lozano Blesa, Zaragoza
  - H. Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link: https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-Interventional, cross-sectional study to describe NOACs management in elderly patients with non-valvular atrial fibrillation (NVAF) in Spain. RE-BELD Study.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the study. Study visit was a routine visit, one of those visits already scheduled in order to follow up the patients' NVAF (Non-Valvular Atrial Fibrillation). Patients were considered included when they agreed to participate in the study and signed the informed consent form.
Groups:
- Dabigatran: Patients in this arm were on treatment with dabigatran (either were receiving 110 milligram (mg) dabigatran twice daily (BID) or 150 mg dabigatran BID) at the time of study visit for their non-valvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC), and had initiated treatment with non-vitamin K antagonist oral anticoagulant (NOAC) at least 3 months before the study visit.
- Rivaroxaban: Patients in this arm were on treatment with rivaroxaban (either were receiving 15 milligram (mg) rivaroxaban once daily (QD) or 20 mg rivaroxaban QD) at the time of study visit for their non-valvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC), and had initiated treatment with non-vitamin K antagonist oral anticoagulant (NOAC) at least 3 months before the study visit.
- Apixaban: Patients in this arm were on treatment with Apixaban (either were receiving 2.5 milligram (mg) apixaban twice daily (BID) or 5 mg apixaban BID) at the time of study visit for their non-valvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC), and had initiated treatment with non-vitamin K antagonist oral anticoagulant (NOAC) at least 3 months before the study visit.
- Edoxaban: Patients in this arm were on treatment with Edoxaban (either were receiving 30 milligram (mg) edoxaban once daily (QD) or 60 mg edoxaban QD) at the time of study visit for their non-valvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC), and had initiated treatment with non-vitamin K antagonist oral anticoagulant (NOAC) at least 3 months before the study visit.
Period: Overall Study
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Started | 192 | 76 | 166 | 66
Completed | 192 | 76 | 166 | 66
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. This is equivalent to the "eligible patients" in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total
Number analyzed (Participants) | 192 | 76 | 166 | 66 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.83 (4.50) | 80.89 (4.64) | 82.29 (4.90) | 82.02 (4.80) | 81.48 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 46 | 94 | 33 | 250
  Male | 115 | 30 | 72 | 33 | 250
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (Kg) [Mean (Standard Deviation); unit: Kilogram (kg)] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Kilogram (kg)
    number analyzed (Participants) | 143 | 70 | 155 | 63 | 431
    (all) | 76.33 (11.53) | 73.23 (13.57) | 74.63 (13.40) | 71.59 (12.41) | 74.52 (12.75)
Weight categorical [Count of Participants; unit: Participants] — Weight was categorized in two categories according to dose adjustment criteria in Non Antagonist of Vitamin K Oral Anticoagulant (NOAC):
  * ≤60 kilograms (kg)
  * >60 kg Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 143 | 70 | 155 | 63 | 431
    ≤60 kg | 13 | 12 | 23 | 14 | 62
    >60 kg | 130 | 58 | 132 | 49 | 369
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  centimeter (cm)
    number analyzed (Participants) | 128 | 68 | 138 | 45 | 379
    (all) | 163.86 (8.28) | 160.88 (8.88) | 162.64 (9.61) | 162.93 (7.75) | 162.77 (8.86)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)] — The formula to obtain Body Mass Index (BMI) of each patient was the following: BMI= kilogram/meter^2 (kg/ m2) = weight (kg)/ height2 (m).
  Mean and Standard Deviation of the BMI for each arm is reported. Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  kilogram/meter^2 (kg/m^2)
    number analyzed (Participants) | 127 | 67 | 136 | 44 | 374
    (all) | 28.58 (4.06) | 28.13 (4.77) | 28.32 (4.71) | 27.46 (3.88) | 28.27 (4.42)
Body mass index categorical (BMI cat) [Count of Participants; unit: Participants] — BMI was categorized in 5 categories, according to the World Health Organization (WHO):
  Underweight: BMI< 18.5 kg/m2 ; Normal weight: 18.5 kg m2 ≤ BMI ≤ 25 kg/m2; Overweight: 25 kg/m2 < BMI ≤ 30 kg/m2; Obese: 30 kg/m2 < BMI ≤ 35 kg/m2; Severely Obese: BMI > 35 kg/m2; Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 127 | 67 | 136 | 44 | 374
    Underweight: BMI< 18.5 kg/m2 | 0 | 0 | 0 | 0 | 0
    Normal weight: 18.5 kg m2≤ BMI≤ 25 kg/m2 | 25 | 16 | 36 | 12 | 89
    Overweight: 25 kg/m2< BMI≤ 30 kg/m2 | 61 | 31 | 55 | 21 | 168
    Obese: 30 kg/m2<BMI≤ 35 kg/m2 | 33 | 17 | 33 | 9 | 92
    Severely Obese: BMI> 35 kg/m2 | 8 | 3 | 12 | 2 | 25
Caregiver [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 169 | 71 | 160 | 63 | 463
    No | 93 | 41 | 78 | 39 | 251
    Yes | 76 | 30 | 82 | 24 | 212
Place where patient is living [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 187 | 72 | 164 | 66 | 489
    Home alone | 17 | 19 | 23 | 10 | 69
    At home with partner/other family member/a friend | 147 | 52 | 119 | 45 | 363
    Other's home (e.g. family member's) | 15 | 1 | 17 | 9 | 42
    Nursing home | 8 | 0 | 5 | 2 | 15
Smoking habit [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 183 | 75 | 163 | 65 | 486
    Ex-smoker | 66 | 17 | 43 | 19 | 145
    Smoker | 6 | 1 | 4 | 1 | 12
    Non-smoker | 111 | 57 | 116 | 45 | 329
Alcohol consumption [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
  Participants
    number analyzed (Participants) | 168 | 72 | 148 | 60 | 448
    Casual or non-consumer | 149 | 66 | 134 | 56 | 405
    Habitual | 19 | 6 | 13 | 3 | 41
    Abuse | 0 | 0 | 1 | 1 | 2
    Dependence | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and Current NOAC Dose According to Sex
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the time of study visit according to sex is reported.
Time Frame: At the single study visit (Day 1).
Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Sex: Male: This arm included all male patients who participated in the study and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Sex: Female: This arm included all female patients who participated in the study and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Sex: Male | Sex: Female
Number analyzed (Participants) | 250 | 250
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 115 | 77
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 30 | 46
  Current NOAC: Apixaban (2.5 mg BID and 5 mg BID patients) | 72 | 94
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 33 | 33
  Dabigatran 110 mg BID: number analyzed (Participants) | 115 | 77
  Dabigatran 110 mg BID | 56 | 41
  Dabigatran 150 mg BID: number analyzed (Participants) | 115 | 77
  Dabigatran 150 mg BID | 59 | 36
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 30 | 46
  Rivaroxaban 15 mg QD | 8 | 23
  Rivaroxaban 20 mg QD: number analyzed (Participants) | 30 | 46
  Rivaroxaban 20 mg QD | 22 | 23
  Apixaban 2.5 mg BID: number analyzed (Participants) | 72 | 94
  Apixaban 2.5 mg BID | 31 | 43
  Apixaban 5 mg BID: number analyzed (Participants) | 72 | 94
  Apixaban 5 mg BID | 41 | 51
  Edoxaban 30 mg QD: number analyzed (Participants) | 33 | 33
  Edoxaban 30 mg QD | 13 | 18
  Edoxaban 60 mg QD: number analyzed (Participants) | 33 | 33
  Edoxaban 60 mg QD | 20 | 15

2. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to Sex
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to sex is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Sex: Male | Sex: Female
Number analyzed (Participants) | 250 | 250
Years | 2.43 (2.19) | 2.22 (1.83)

3. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and NOAC Dose According to Age (Categorical)
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the time of study visit according to patients' age is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Age: 75-79 Years: This arm included all patients aged between 75-79 years who participated in the study and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Age: 80-84 Years: This arm included all patients aged between 80-84 years who participated in the study and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Age: ≥85 Years: This arm included all patients ≥85 years old who participated in the study and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Age: 75-79 Years | Age: 80-84 Years | Age: ≥85 Years
Number analyzed (Participants) | 210 | 152 | 138
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 93 | 59 | 40
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 34 | 23 | 19
  Current NOAC: Apixaban (2.5 mg BID and 5 mg BID patients) | 59 | 48 | 59
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 24 | 22 | 20
  Dabigatran 110 mg BID: number analyzed (Participants) | 93 | 59 | 40
  Dabigatran 110 mg BID | 22 | 39 | 36
  Dabigatran 150 mg BID: number analyzed (Participants) | 93 | 59 | 40
  Dabigatran 150 mg BID | 71 | 20 | 4
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 34 | 23 | 19
  Rivaroxaban 15 mg QD | 10 | 9 | 12
  Rivaroxaban 20 mg QD: number analyzed (Participants) | 34 | 23 | 19
  Rivaroxaban 20 mg QD | 24 | 14 | 7
  Apixaban 2.5 mg BID: number analyzed (Participants) | 59 | 48 | 59
  Apixaban 2.5 mg BID | 16 | 21 | 37
  Apixaban 5 mg BID: number analyzed (Participants) | 59 | 48 | 59
  Apixaban 5 mg BID | 43 | 27 | 22
  Edoxaban 30 mg QD: number analyzed (Participants) | 24 | 22 | 20
  Edoxaban 30 mg QD | 7 | 11 | 13
  Edoxaban 60 mg QD: number analyzed (Participants) | 24 | 22 | 20
  Edoxaban 60 mg QD | 17 | 11 | 7

4. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to Patient's Age (Categorical)
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to patient's age (categorical) is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Age: 75-79 Years | Age: 80-84 Years | Age: ≥85 Years
Number analyzed (Participants) | 210 | 152 | 138
Years | 2.33 (2.07) | 2.32 (1.93) | 2.32 (2.05)

5. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and NOAC Dose According to a Prior Diagnosis of Heart Failure
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the time of study visit according to a prior diagnosis of heart failure is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Heart Failure: No: This arm included patients who participated in the study and had no prior diagnosis of heart failure and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Heart Failure: Yes: This arm included patients who participated in the study and had prior diagnosis of heart failure and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Heart Failure: No | Heart Failure: Yes
Number analyzed (Participants) | 316 | 184
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 129 | 63
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 54 | 22
  Current NOAC: Apixaban (2.5 mg BID and 5 mg patients) | 96 | 70
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 37 | 29
  Dabigatran 110 mg BID: number analyzed (Participants) | 129 | 63
  Dabigatran 110 mg BID | 63 | 34
  Dabigatran 150 mg BID: number analyzed (Participants) | 129 | 63
  Dabigatran 150 mg BID | 66 | 29
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 54 | 22
  Rivaroxaban 15 mg QD | 21 | 10
  Rivaroxaban 20 mg QD: number analyzed (Participants) | 54 | 22
  Rivaroxaban 20 mg QD | 33 | 12
  Apixaban 2.5 mg BID: number analyzed (Participants) | 96 | 70
  Apixaban 2.5 mg BID | 31 | 43
  Apixaban 5 mg BID: number analyzed (Participants) | 96 | 70
  Apixaban 5 mg BID | 65 | 27
  Edoxaban 30 mg QD: number analyzed (Participants) | 37 | 29
  Edoxaban 30 mg QD | 16 | 15
  Edoxaban 60 mg QD: number analyzed (Participants) | 37 | 29
  Edoxaban 60 mg QD | 21 | 14

6. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to a Prior Diagnosis of Heart Failure
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to a prior diagnosis of heart failure is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Heart Failure: No | Heart Failure: Yes
Number analyzed (Participants) | 316 | 184
Years | 2.27 (2.02) | 2.41 (2.02)

7. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and NOAC Dose According to Coronary Artery Disease
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the study visit according to patients' coronary artery disease is reported.
Time Frame: At the single study visit (Day 1).
Population: Full Analysis Set (FAS): All enrolled subjects who provided informed consent for this study and fulfilled all selection criteria. Only participants with non-missing outcomes were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Disease: No: This arm included patients who participated in the study and had no coronary artery disease and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Coronary Artery Disease: Yes: This arm included patients who participated in the study and had coronary artery disease and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Coronary Artery Disease: No | Coronary Artery Disease: Yes
Number analyzed (Participants) | 414 | 82
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 156 | 35
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 63 | 13
  Current NOAC: Apixaban (2.5 mg BID and 5 mg BID patients) | 142 | 21
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 53 | 13
  Dabigatran 110 mg BID: number analyzed (Participants) | 156 | 35
  Dabigatran 110 mg BID | 78 | 19
  Dabigatran 150 mg BID: number analyzed (Participants) | 156 | 35
  Dabigatran 150 mg BID | 78 | 16
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 63 | 13
  Rivaroxaban 15 mg QD | 23 | 8
  Rivaroxaban 20 mg QD: number analyzed (Participants) | 63 | 13
  Rivaroxaban 20 mg QD | 40 | 5
  Apixaban 2.5 mg BID: number analyzed (Participants) | 142 | 21
  Apixaban 2.5 mg BID | 62 | 10
  Apixaban 5 mg BID: number analyzed (Participants) | 142 | 21
  Apixaban 5 mg BID | 80 | 11
  Edoxaban 30 mg QD: number analyzed (Participants) | 53 | 13
  Edoxaban 30 mg QD | 23 | 8
  Edoxaban 60 mg QD: number analyzed (Participants) | 53 | 13
  Edoxaban 60 mg QD | 30 | 5

8. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to Coronary Artery Disease
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to patients' coronary artery disease is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Coronary Artery Disease: No | Coronary Artery Disease: Yes
Number analyzed (Participants) | 414 | 82
Years | 2.38 (2.02) | 2.04 (1.99)

9. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and NOAC Dose According to Diabetes
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the time of study visit according to patients' diabetes is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Diabetes: No: This arm included patients who participated in the study and had no diabetes were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Diabetes: Yes: This arm included patients who participated in the study and had diabetes and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Diabetes: No | Diabetes: Yes
Number analyzed (Participants) | 346 | 154
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 135 | 57
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 51 | 25
  Current NOAC: Apixaban (2.5 mg BID and 5 mg BID patients) | 113 | 53
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 47 | 19
  Dabigatran 110 mg BID: number analyzed (Participants) | 135 | 57
  Dabigatran 110 mg BID | 68 | 29
  Dabigatran 150 mg BID: number analyzed (Participants) | 135 | 57
  Dabigatran 150 mg BID | 67 | 28
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 51 | 25
  Rivaroxaban 15 mg QD | 22 | 9
  Rivaroxaban 20 mg QD: number analyzed (Participants) | 51 | 25
  Rivaroxaban 20 mg QD | 29 | 16
  Apixaban 2.5 mg BID: number analyzed (Participants) | 113 | 53
  Apixaban 2.5 mg BID | 51 | 23
  Apixaban 5 mg BID: number analyzed (Participants) | 113 | 53
  Apixaban 5 mg BID | 62 | 30
  Edoxaban 30 mg QD: number analyzed (Participants) | 47 | 19
  Edoxaban 30 mg QD | 21 | 10
  Edoxaban 60 mg QD: number analyzed (Participants) | 47 | 19
  Edoxaban 60 mg QD | 26 | 9

10. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to Diabetes
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to patients' diabetes is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Diabetes: No | Diabetes: Yes
Number analyzed (Participants) | 346 | 154
Years | 2.39 (2.00) | 2.17 (2.07)

11. Primary Outcome: Type of Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and NOAC Dose According to Chronic Kidney Disease
Description: Number of patients receiving dabigatran (Current NOAC: Dabigatran), rivaroxaban (Current NOAC: Rivaroxaban), apixaban (Current NOAC: Apixaban), edoxaban (Current NOAC: Edoxaban), dabigatran 110 mg (twice daily) BID, dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD at the time of study visit according to patients' chronic kidney disease is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Chronic Kidney Disease: No: This arm included patients who participated in the study and had no chronic kidney disease were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
- Chronic Kidney Disease: Yes: This arm included patients who participated in the study and had chronic kidney disease and were receiving any Non-vitamin K antagonist oral anticoagulant (NOAC) (either dabigatran, rivaroxaban, apixaban or edoxaban) for their nonvalvular atrial fibrillation (NVAF), according to the indication approved in their Summary of Product Characteristics (SmPC).
Arm/Group | Chronic Kidney Disease: No | Chronic Kidney Disease: Yes
Number analyzed (Participants) | 408 | 92
Participants
  Current NOAC: Dabigatran (110 mg BID and 150 mg BID patients) | 166 | 26
  Current NOAC: Rivaroxaban (15 mg QD and 20 mg QD patients) | 64 | 12
  Current NOAC: Apixaban (2.5 mg BID and 5 mg BID patients) | 130 | 36
  Current NOAC: Edoxaban (30 mg QD and 60 mg QD patients) | 48 | 18
  Dabigatran 110 mg BID: number analyzed (Participants) | 166 | 26
  Dabigatran 110 mg BID | 76 | 21
  Dabigatran 150 mg BID: number analyzed (Participants) | 166 | 26
  Dabigatran 150 mg BID | 90 | 5
  Rivaroxaban 15 mg QD: number analyzed (Participants) | 64 | 12
  Rivaroxaban 15 mg QD | 19 | 12
  Rivaroxaban 20mg QD: number analyzed (Participants) | 64 | 12
  Rivaroxaban 20mg QD | 45 | 0
  Apixaban 2.5 mg BID: number analyzed (Participants) | 130 | 36
  Apixaban 2.5 mg BID | 43 | 31
  Apixaban 5 mg BID: number analyzed (Participants) | 130 | 36
  Apixaban 5 mg BID | 87 | 5
  Edoxaban 30 mg QD: number analyzed (Participants) | 48 | 18
  Edoxaban 30 mg QD | 17 | 14
  Edoxaban 60 mg QD: number analyzed (Participants) | 48 | 18
  Edoxaban 60 mg QD | 31 | 4

12. Primary Outcome: Number of Years Since First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation to Study Visit According to Chronic Kidney Disease
Description: Number of years since first Non-vitamin K antagonist oral anticoagulant (NOAC) initiation to study visit according to patients' chronic kidney disease is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Chronic Kidney Disease: No | Chronic Kidney Disease: Yes
Number analyzed (Participants) | 408 | 92
Years | 2.34 (2.05) | 2.25 (1.89)

13. Secondary Outcome: Serum Creatinine Concentration From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Serum creatinine concentration from the last available blood sample analysis was retrieved from patients' medical records. Serum creatinine concentration from the last available blood sample analysis according to current NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dl)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 159 | 63 | 122 | 47
milligram/deciliter (mg/dl) | 1.00 (0.23) | 1.05 (0.29) | 1.15 (0.41) | 1.14 (0.39)

14. Secondary Outcome: Creatinine Clearance From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients' medical records were used to retrieve the creatinine clearance (CrCl). These results were directly collected in the Electronic Case Report Form (eCRF).
  In cases where CrCl was not available in patients's medical record but serum creatinine was available, CrCl was estimated using Cockcroft-Gault formula:
  CrCl = (140 - Age(years)) x Weight (kilogram) x [0.85 if female] / 72 x [Serum Creatinine (milligram/deciliterL)]
  Reported are Crcl values which are calculated according to:
  * Cockcroft-Gault formula and CrCl values directly collected in the eCRF
  * Cockcroft-Gault formula only
  * Directly collected in the eCRF
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter/minute (ml/min)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 141 | 71 | 156 | 46
milliliter/minute (ml/min)
  CrCl calculated by Cockcroft-Gault formula and CrCl values directly collected in the eCRF | 63.50 (18.49) | 55.42 (17.59) | 54.45 (18.65) | 53.04 (18.40)
  Calculated by Cockcroft-Gault formula only: number analyzed (Participants) | 110 | 60 | 114 | 46
  Calculated by Cockcroft-Gault formula only | 62.72 (18.82) | 54.59 (17.79) | 53.77 (19.35) | 52.83 (18.84)
  Directly collected in the eCRF: number analyzed (Participants) | 31 | 11 | 42 | 17
  Directly collected in the eCRF | 66.27 (17.27) | 59.98 (16.47) | 56.30 (16.69) | 53.59 (17.69)

15. Secondary Outcome: Number of Participants in Each Category of Creatinine Clearance Range From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients' medical records were used to retrieve the creatinine clearance (CrCl). These results were directly collected in the Electronic Case Report Form (eCRF).
  In cases where CrCl was not available in patients' medical record but serum creatinine was available, CrCl was estimated using Cockcroft-Gault formula:
  CrCl = (140 - Age(years)) x Weight (kilogram) x [0.85 if female] / 72 x [Serum Creatinine (milligram/deciliterL)]
  The number of participants for each of the following creatinine clearance (CrCl) ranges is reported:
  * CrCl ≥90: Kidney damage with normal or increased glomerular filtration rate (GFR)
  * CrCl 60-89: Kidney damage with mild decreased GFR
  * CrCl 30-59: Moderate decrease in GFR
  * CrCl 15-29: Severe decrease in GFR
  * CrCl <15: Kidney failure
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 141 | 71 | 156 | 63
Participants
  <15 ml/min/1.73m^2 | 0 | 0 | 0 | 0
  15-29 ml/min/1.73m^2 | 0 | 3 | 10 | 7
  30-59 ml/min/1.73m^2 | 72 | 41 | 92 | 37
  60-89 ml/min/1.73m^2 | 55 | 25 | 46 | 18
  ≥90 ml/min/1.73m^2 | 14 | 2 | 8 | 1

16. Secondary Outcome: Aspartate Aminotransferase (AST) Concentration From the Last Available Blood Sample According to Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients' medical records were used to retrieve AST concentration. AST concentration from the last available blood sample according to non-vitamin K antagonist oral anticoagulant (NOAC) type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 128 | 62 | 138 | 59
international units per liter (IU/L) | 24.13 (11.34) | 21.60 (7.43) | 25.57 (16.01) | 20.81 (8.58)

17. Secondary Outcome: Alanine Aminotransferase (ALT) From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients's medical records were used to retrieve ALT concentration. ALT concentration from the last available blood sample according to NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units per liter (UI/L)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 127 | 66 | 143 | 62
units per liter (UI/L) | 22.38 (13.66) | 18.28 (8.95) | 21.52 (17.81) | 20.15 (20.76)

18. Secondary Outcome: Bilirubin Concentration From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients's medical records were used to retrieve bilirubin concentration. Bilirubin concentration from the last available blood sample according to NOAC type is reported.Results from the last available blood sample analysis from patients' medical records were used to retrieve bilirubin concentration. Bilirubin concentration from the last available blood sample according to NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dl)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 103 | 53 | 119 | 45
milligram/deciliter (mg/dl) | 0.83 (0.47) | 0.79 (0.51) | 0.74 (0.47) | 0.75 (0.37)

19. Secondary Outcome: Haemoglobin Concentration From the Last Available Blood Sample According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients' medical records were used to retrieve haemoglobin concentration. Haemoglobin concentration from the last available blood sample according to NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dl)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 181 | 75 | 165 | 64
gram/deciliter (g/dl) | 13.23 (1.66) | 13.37 (1.61) | 12.99 (1.90) | 13.17 (1.92)

20. Secondary Outcome: Platelet Levels From the Last Available Blood Sample According to Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Results from the last available blood sample analysis from patients's medical records were used to retrieve platelet levels. Platelet levels from the last available blood sample according to NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: x 10^3/microliter (μL)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 174 | 73 | 160 | 64
x 10^3/microliter (μL) | 203.37 (60.50) | 222.07 (77.13) | 215.59 (81.48) | 189.45 (68.80)

21. Secondary Outcome: Number of Patients in Each Category of Serum Creatinine, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Bilirubin, Hemoglobin and Platelet Levels According to Current Non-vitamin K Antagonist Oral (NOAC) Type
Description: Results from the last available blood sample analysis from patients' medical records were used to retrieve serum creatinine, ALT, AST, bilirubin, hemoglobin concentration and platelet levels.
  For each reported laboratory parameter the values were categorized in two categories:
  Serum creatinine:
  * Normal value : 0.6-1.2 mg/dl in males and 0.5-1.1 mg/dl in females
  * High/low value
  ALT:
  * Normal values: 7-55 units per liter (UI/L)
  * High/low values
  AST:
  * Normal values: 8-48 UI/L
  * High/low values
  Bilirubin:
  * Normal values: 0.2-1.2 milligram per deciliter (mg/dl)
  * High/low values
  Haemoglobin:
  * Normal values: 12-18 gram/deciliter (g/dL)
  * High/low values
  Platelets:
  * Normal values: 150-450 x10^3/µL
  * High/low values
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Serum creatinine: number analyzed (Participants) | 159 | 63 | 122 | 47
  Serum creatinine: Normal levels | 132 | 44 | 72 | 32
  Serum creatinine: High/low levels | 27 | 19 | 50 | 15
  AST: number analyzed (Participants) | 128 | 62 | 138 | 59
  AST: Normal levels | 122 | 61 | 127 | 59
  AST: High/low levels | 6 | 1 | 11 | 0
  ALT: number analyzed (Participants) | 127 | 66 | 143 | 62
  ALT: Normal levels | 121 | 65 | 133 | 59
  ALT: High/low levels | 6 | 1 | 10 | 3
  Total bilirubin: number analyzed (Participants) | 103 | 53 | 119 | 45
  Total bilirubin: Normal levels | 91 | 46 | 109 | 41
  Total bilirubin: High/low levels | 12 | 7 | 10 | 4
  Hemoglobin: number analyzed (Participants) | 181 | 75 | 165 | 64
  Hemoglobin: Normal levels | 143 | 63 | 121 | 50
  Hemoglobin: High/low levels | 38 | 12 | 44 | 14
  Platelet: number analyzed (Participants) | 174 | 73 | 160 | 64
  Platelet: Normal levels | 140 | 65 | 128 | 48
  Platelet: High/low levels | 34 | 8 | 32 | 16

22. Secondary Outcome: Non-valvular Atrial Fibrillation (NVAF) Characteristics: Number of Years Since NVAF Diagnosis According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The number of years since NVAF diagnosis was obtained from number of years between date of NVAF diagnosis and date of study visit.
  The date of NVAF diagnosis was retrieved from patient's medical records. The number of years since NVAF diagnosis and date of study visit is reported for:
  * All patients;
  * Patients treated previously with vitamin K antagonists (VKA);
  * Patients treated with NOAC as first anticoagulant .
Time Frame: At the single study visit (day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 165 | 66
Years
  All patients | 4.78 (4.26) | 5.85 (4.70) | 6.01 (6.54) | 5.63 (4.99)
  Patients treated previously with VKA: number analyzed (Participants) | 109 | 40 | 93 | 44
  Patients treated previously with VKA | 6.30 (4.59) | 7.95 (4.87) | 7.60 (5.43) | 7.59 (4.94)
  Patients treated with NOAC as first anticoagulant: number analyzed (Participants) | 83 | 36 | 72 | 22
  Patients treated with NOAC as first anticoagulant | 2.79 (2.71) | 3.52 (3.21) | 3.95 (7.28) | 1.72 (1.74)

23. Secondary Outcome: Non-valvular Atrial Fibrillation (NVAF) Characteristics: Number of Patients in Each Category of NVAF Type According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: NVAF was categorized in four categories:
  * Persistent;
  * Long standing persistent;
  * Permanent;
  * Paroxysmal.
Time Frame: At the single study visit (day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 189 | 71 | 160 | 63
Participants
  Persistent | 32 | 11 | 31 | 12
  Long standing persistent | 21 | 3 | 10 | 5
  Permanent | 99 | 26 | 66 | 36
  Paroxysmal | 37 | 31 | 53 | 10

24. Secondary Outcome: Non-valvular Atrial Fibrillation (NVAF) Characteristics: Number of Patients in Each Category of EHRA Scale for Atrial Fibrillation (AF) Related Symptoms According to Current NOAC Type
Description: The European Heart Rhythm Association (EHRA) score of atrial fibrillation is a classification system for the extent of atrial fibrillation. It places patients in one of five categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  The EHRA categories are the following:
  1-no symptoms 2a-mild symptoms; normal daily activity not affected. 2b-moderate symptoms; normal daily activity not affected. 3-severe symptoms; normal daily activity affected. 4-disabling; normal daily activity discontinued.
Time Frame: At the single study visit (day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 188 | 69 | 157 | 62
Participants
  1-none | 47 | 25 | 52 | 17
  2a-mild | 83 | 30 | 70 | 31
  2b-moderate | 45 | 11 | 28 | 11
  3-severe | 10 | 3 | 6 | 3
  4-disabling | 3 | 0 | 1 | 0

25. Secondary Outcome: Number of Patients in Each Category of Cardioversion, Ablation, Coronary Interventions and Pacemaker Carrier According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Number of patients with (category Yes) and without (category No) cardioversion, ablation, coronary interventions and pacemaker carrier according to current NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Cardioversion: number analyzed (Participants) | 187 | 76 | 165 | 66
  Cardioversion: No | 171 | 70 | 151 | 57
  Cardioversion: Yes | 16 | 6 | 14 | 9
  Ablation: number analyzed (Participants) | 189 | 76 | 166 | 66
  Ablation: No | 178 | 75 | 160 | 64
  Ablation: Yes | 11 | 1 | 6 | 2
  Coronary interventions: number analyzed (Participants) | 189 | 76 | 165 | 65
  Coronary interventions: No | 167 | 65 | 148 | 60
  Coronary interventions: Yes | 22 | 11 | 17 | 5
  Pacemaker carrier: number analyzed (Participants) | 189 | 76 | 166 | 66
  Pacemaker carrier: No | 166 | 67 | 151 | 58
  Pacemaker carrier: Yes | 23 | 9 | 15 | 8

26. Secondary Outcome: Number of Patients in Each Category of Coronary Interventions According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Number of patients in each category of coronary interventions according to current non-vitamin K antagonist oral anticoagulant (NOAC) type is reported.
  Coronary interventions were categorized in:
  * Percutaneous coronary intervention and
  * Coronary artery bypass grafting.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who underwent coronary interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 22 | 11 | 17 | 5
Participants
  Percutaneous coronary intervention | 19 | 9 | 14 | 4
  Coronary artery bypass grafting | 3 | 2 | 3 | 1

27. Secondary Outcome: Clinical Risk Factors: Number of Patients in Each Category of Heart Failure, Coronary Artery Disease, Sleep Apnoea-hypopnoea Syndrome, Hypertension and Hyperlipidaemia According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Number of patients in each category of heart failure, coronary artery disease, sleep apnoea-hypopnoea syndrome, hypertension and hyperlipidaemia according to current non-vitamin K antagonist oral anticoagulant (NOAC) type is reported.
  Heart failure, coronary artery disease, sleep apnoea-hypopnoea syndrome, hypertension and hyperlipidaemia were categorized in the following two categories:
  * No;
  * Yes.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Heart failure: No | 129 | 54 | 96 | 37
  Heart failure: Yes | 63 | 22 | 70 | 29
  Coronary artery disease: number analyzed (Participants) | 191 | 76 | 163 | 66
  Coronary artery disease: No | 156 | 63 | 142 | 53
  Coronary artery disease: Yes | 35 | 13 | 21 | 13
  Sleep apnoea-hypopnoea syndrome: number analyzed (Participants) | 189 | 76 | 163 | 66
  Sleep apnoea-hypopnoea syndrome: No | 170 | 70 | 152 | 57
  Sleep apnoea-hypopnoea syndrome: Yes | 19 | 6 | 11 | 9
  Hypertension: No | 46 | 13 | 22 | 7
  Hypertension: Yes | 146 | 63 | 144 | 59
  Hyperlipidaemia: number analyzed (Participants) | 192 | 76 | 165 | 66
  Hyperlipidaemia: No | 76 | 28 | 68 | 17
  Hyperlipidaemia: Yes | 116 | 48 | 97 | 49

28. Secondary Outcome: Clinical Risk Factors: Number of Heart Failure Patients in Each Category of New York Heart Association (NYHA) Classification According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The NYHA provides a simple way of classifying the extent of heart failure and it has 4 categories:
  * A - No objective evidence of cardiovascular disease
  * B - Objective evidence of minimal cardiovascular disease
  * C - Objective evidence of moderately severe cardiovascular disease
  * D - Objective evidence of severe cardiovascular disease Number of heart failure patients in each category of New York Heart Association (NYHA) classification according to current NOAC type is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS with heart failure. NYHA classification for heart failure patients is missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 61 | 20 | 61 | 22
Participants
  A - No objective evidence of cardiovascular disease | 2 | 0 | 3 | 0
  B - Objective evidence of minimal cardiovascular disease | 39 | 12 | 25 | 8
  C - Objective evidence of moderately severe cardiovascular disease | 18 | 6 | 29 | 12
  D - Objective evidence of severe cardiovascular disease | 2 | 2 | 4 | 2

29. Secondary Outcome: Clinical Risk Factors: Left Ventricular Ejection Fraction According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Left ventricular ejection fraction (LVEF) according to current non-vitamin K antagonist oral anticoagulant (NOAC) type is reported. LVEF was obtained from the patients' medical records.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent ejection fraction (%)
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 181 | 58 | 130 | 57
percent ejection fraction (%) | 59.47 (9.66) | 59.43 (10.45) | 58.85 (12.27) | 57.91 (12.57)

30. Secondary Outcome: Age-adjusted Charlson Comorbidity Index Score According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. Up to 12 comorbidities with various weightings can result in a maximum score of 24. The minimum score is zero.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 75 | 165 | 66
Score on a scale | 5.26 (1.74) | 5.39 (1.63) | 5.99 (2.04) | 6.27 (2.41)

31. Secondary Outcome: Number of Patients With and Without the Comorbidities Included in the Charlson Comorbidity Index According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Number of patients with (Yes) and without (No) the comorbidities which were included in the Charlson Comorbidity Index according to current NOAC type is reported.
  The comorbidities which were included in the Charlson Comorbidity Index were the following:
  * Myocardial infarction
  * Congestive heart failure
  * Peripheral vascular disease
  * Cerebrovascular disease
  * Dementia
  * Chronic Obstructive Pulmonary Disease (COPD)
  * Connective tissue disease
  * Peptic ulcer disease
  * Liver disease (No/Mild/Moderate to severe)
  * Diabetes mellitus (No/Uncomplicated/End-organ damage)
  * Hemiplegia
  * Moderate to severe renal disease
  * Solid Tumor (No/Localized/Metastatic)
  * Leukaemia
  * Lymphoma
  * Acquired Immune Deficiency Syndrome (AIDS).
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Myocardial infarction; No: number analyzed (Participants) | 192 | 76 | 165 | 66
  Myocardial infarction; No | 176 | 65 | 147 | 55
  Myocardial infarction; Yes: number analyzed (Participants) | 192 | 76 | 165 | 66
  Myocardial infarction; Yes | 16 | 11 | 18 | 11
  Congestive heart failure: No | 129 | 55 | 96 | 38
  Congestive heart failure: Yes | 63 | 21 | 70 | 28
  Peripheral vascular disease: No: number analyzed (Participants) | 192 | 75 | 166 | 66
  Peripheral vascular disease: No | 172 | 70 | 151 | 59
  Peripheral vascular disease: Yes: number analyzed (Participants) | 192 | 75 | 166 | 66
  Peripheral vascular disease: Yes | 20 | 5 | 15 | 7
  Cerebrovascular disease: No | 153 | 63 | 133 | 57
  Cerebrovascular disease: Yes | 39 | 13 | 33 | 9
  Dementia: No | 188 | 72 | 153 | 60
  Dementia: Yes | 4 | 4 | 13 | 6
  COPD: No: number analyzed (Participants) | 192 | 76 | 165 | 66
  COPD: No | 161 | 66 | 141 | 54
  COPD: Yes: number analyzed (Participants) | 192 | 76 | 165 | 66
  COPD: Yes | 31 | 10 | 24 | 12
  Connective tissue disease: No | 189 | 76 | 164 | 66
  Connective tissue disease: Yes | 3 | 0 | 2 | 0
  Peptic ulcer disease: No | 187 | 74 | 156 | 65
  Peptic ulcer disease: Yes | 5 | 2 | 10 | 1
  Liver disease: No | 190 | 74 | 161 | 65
  Liver disease: Mild | 2 | 2 | 5 | 1
  Liver disease: Moderate to severe | 0 | 0 | 0 | 0
  Diabetes mellitus: No | 135 | 51 | 113 | 47
  Diabetes mellitus: Uncomplicated | 48 | 18 | 36 | 11
  Diabetes mellitus: End-organ damage | 9 | 7 | 17 | 8
  Hemiplegia: No | 191 | 76 | 164 | 62
  Hemiplegia: Yes | 1 | 0 | 2 | 4
  Moderate to severe renal disease: No | 166 | 64 | 130 | 48
  Moderate to severe renal disease: Yes | 26 | 12 | 36 | 18
  Solid tumor: No | 178 | 69 | 148 | 57
  Solid tumor: Localized | 13 | 7 | 16 | 7
  Solid tumor: Metastatic | 1 | 0 | 2 | 2
  Leukaemia: No | 192 | 76 | 166 | 66
  Leukaemia: Yes | 0 | 0 | 0 | 0
  Lymphoma: No | 192 | 74 | 165 | 65
  Lymphoma: Yes | 0 | 2 | 1 | 1
  AIDS: No | 192 | 76 | 165 | 66
  AIDS: Yes | 0 | 0 | 1 | 0

32. Secondary Outcome: Number of Patients With and Without Any History of Thromboembolic Events, Number of Patients in Each Category of Different Types of Thromboembolic Events According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Reported is the number of patients in each category of:
  * Any history of thromboembolic events
  * Transient Ischemic Attack (TIA)
  * Ischemic stroke
  * Haemorrhagic stroke
  * Embolism systemic
  * Deep vein thrombosis
  * Pulmonary embolism.
  Any history of thromboembolic events, Transient Ischemic Attack (TIA), ischemic stroke, haemorrhagic stroke, embolism systemic, deep vein thrombosis and pulmonary embolism were categorized in the following two categories:
  * No
  * Yes.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Any history of thromboembolic events: No | 153 | 53 | 120 | 48
  Any history of thromboembolic events: Yes | 39 | 23 | 46 | 18
  Transient Ischemic Attack (TIA): number analyzed (Participants) | 190 | 75 | 163 | 66
  Transient Ischemic Attack (TIA): No | 180 | 66 | 155 | 64
  Transient Ischemic Attack (TIA): Yes | 10 | 9 | 8 | 2
  Ischemic stroke: number analyzed (Participants) | 192 | 72 | 166 | 65
  Ischemic stroke: No | 173 | 65 | 146 | 60
  Ischemic stroke: Yes | 19 | 7 | 20 | 5
  Haemorrhagic stroke: number analyzed (Participants) | 190 | 73 | 164 | 65
  Haemorrhagic stroke: No | 189 | 73 | 163 | 65
  Haemorrhagic stroke: Yes | 1 | 0 | 1 | 0
  Embolism systemic: number analyzed (Participants) | 191 | 73 | 164 | 65
  Embolism systemic: No | 191 | 73 | 164 | 63
  Embolism systemic: Yes | 0 | 0 | 0 | 2
  Deep vein thrombosis: number analyzed (Participants) | 191 | 73 | 164 | 65
  Deep vein thrombosis: No | 190 | 71 | 162 | 65
  Deep vein thrombosis: Yes | 1 | 2 | 2 | 0
  Pulmonary embolism: number analyzed (Participants) | 191 | 74 | 164 | 65
  Pulmonary embolism: No | 190 | 73 | 161 | 64
  Pulmonary embolism: Yes | 1 | 1 | 3 | 1

33. Secondary Outcome: Number of Patients in Each Category of Stable Angina, Unstable Angina, Myocardial Infarction With ST Segment Elevation and Myocardial Infarction Without ST Segment Elevation According to Current NOAC Type
Description: Number of patients in each category of stable angina, unstable angina, myocardial infarction with ST segment elevation and myocardial infarction without ST segment elevation according to current non-vitamin K antagonist oral anticoagulant (NOAC) type is reported.
  Stable angina, unstable angina, myocardial infarction with ST segment elevation myocardial infarction without ST segment elevation were categorized in the following 2 categories:
  * Yes;
  * No.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Stable angina: number analyzed (Participants) | 191 | 73 | 165 | 65
  Stable angina: No | 187 | 73 | 161 | 64
  Stable angina: Yes | 4 | 0 | 4 | 1
  Unstable angina: number analyzed (Participants) | 191 | 73 | 164 | 65
  Unstable angina: No | 190 | 72 | 158 | 64
  Unstable angina: Yes | 1 | 1 | 6 | 1
  Myocardial infarction with ST segment elevation: number analyzed (Participants) | 191 | 73 | 164 | 65
  Myocardial infarction with ST segment elevation: No | 183 | 65 | 153 | 62
  Myocardial infarction with ST segment elevation: Yes | 8 | 8 | 11 | 3
  Myocardial infarction without ST segment elevation: number analyzed (Participants) | 191 | 73 | 164 | 65
  Myocardial infarction without ST segment elevation: No | 183 | 69 | 156 | 57
  Myocardial infarction without ST segment elevation: Yes | 8 | 4 | 8 | 8

34. Secondary Outcome: Total Number of Thromboembolic Events, Number of Each Type of Thromboembolic Events, Number of Stable and Unstable Anginas, and Number of ST and Non-ST Myocardial Infarction According to Current NOAC Type
Description: Total number of thromboembolic events, number of each type of thromboembolic events, number of stable and unstable anginas, and number of ST and non-ST myocardial infarction according to current non-vitamin K antagonist oral anticoagulant (NOAC) type is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
events
  Total number of thromboembolic events | 0.29 (0.66) | 0.54 (1.24) | 0.49 (1.19) | 0.36 (0.69)
  Number of Transient Ischemic Attack (TIA): number analyzed (Participants) | 190 | 75 | 163 | 63
  Number of Transient Ischemic Attack (TIA) | 0.05 (0.22) | 0.19 (0.63) | 0.06 (0.25) | 0.03 (0.17)
  Number of ischemic strokes: number analyzed (Participants) | 192 | 72 | 166 | 65
  Number of ischemic strokes | 0.10 (0.30) | 0.10 (0.30) | 0.13 (0.35) | 0.09 (0.34)
  Number of haemorrhagic strokes: number analyzed (Participants) | 190 | 73 | 164 | 65
  Number of haemorrhagic strokes | 0.01 (0.07) | 0.00 (0.00) | 0.01 (0.08) | 0.00 (0.00)
  Number of embolism systemic: number analyzed (Participants) | 191 | 73 | 164 | 65
  Number of embolism systemic | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.03 (0.17)
  Number of deep vein thrombosis: number analyzed (Participants) | 191 | 73 | 164 | 65
  Number of deep vein thrombosis | 0.01 (0.14) | 0.05 (0.37) | 0.01 (0.11) | 0.00 (0.00)
  Number of pulmonary embolisms: number analyzed (Participants) | 191 | 74 | 164 | 65
  Number of pulmonary embolisms | 0.01 (0.07) | 0.01 (0.12) | 0.02 (0.13) | 0.02 (0.12)
  Number of stable anginas: number analyzed (Participants) | 191 | 73 | 165 | 65
  Number of stable anginas | 0.02 (0.14) | 0.00 (0.00) | 0.02 (0.15) | 0.02 (0.12)
  Number of unstable anginas: number analyzed (Participants) | 191 | 73 | 164 | 65
  Number of unstable anginas | 0.01 (0.07) | 0.01 (0.12) | 0.12 (0.74) | 0.02 (0.12)
  Number of myocardial infarctions with ST segment elevation | 0.04 (0.20) | 0.12 (0.37) | 0.07 (0.25) | 0.05 (0.21)
  Number of myocardial infarctions without ST segment elevation | 0.05 (0.24) | 0.07 (0.30) | 0.06 (0.29) | 0.12 (0.33)

35. Secondary Outcome: Number of Patients With and Without Any History of Bleeding Events and Number of Patients in Each Category of Bleeding Type According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Number of patients with (category Yes) and without (category No) any history of bleeding events and number of patients in each category of the following bleeding types is reported:
  * Intracranial
  * Digestive
  * Genitourinary
  * Gingival
  * Nasal
  * Pulmonary
  * Articular-muscular
  * Conjunctival.
  Intracranial, digestive, genitourinary, gingival, nasal, pulmonary, articular-muscular, conjunctival were categorized in two categories:
  * No
  * Yes.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Any history of bleeding events: number analyzed (Participants) | 191 | 76 | 166 | 65
  Any history of bleeding events: No | 177 | 68 | 120 | 56
  Any history of bleeding events: Yes | 14 | 8 | 46 | 9
  Intracranial: number analyzed (Participants) | 191 | 76 | 165 | 65
  Intracranial: No | 188 | 74 | 158 | 64
  Intracranial: Yes | 3 | 2 | 7 | 1
  Digestive: number analyzed (Participants) | 191 | 76 | 166 | 65
  Digestive: No | 183 | 73 | 140 | 62
  Digestive: Yes | 8 | 3 | 26 | 3
  Genitourinary: number analyzed (Participants) | 191 | 76 | 164 | 65
  Genitourinary: No | 189 | 76 | 158 | 63
  Genitourinary: Yes | 2 | 0 | 6 | 2
  Gingival: number analyzed (Participants) | 191 | 76 | 165 | 65
  Gingival: No | 191 | 75 | 163 | 64
  Gingival: Yes | 0 | 1 | 2 | 1
  Nasal: number analyzed (Participants) | 191 | 76 | 165 | 65
  Nasal: No | 191 | 76 | 157 | 62
  Nasal: Yes | 0 | 0 | 8 | 3
  Pulmonary: number analyzed (Participants) | 191 | 76 | 165 | 65
  Pulmonary: No | 191 | 76 | 162 | 64
  Pulmonary: Yes | 0 | 0 | 3 | 1
  Articular-muscular: number analyzed (Participants) | 191 | 76 | 165 | 65
  Articular-muscular: No | 189 | 76 | 162 | 65
  Articular-muscular: Yes | 2 | 0 | 3 | 0
  Conjunctival: number analyzed (Participants) | 191 | 76 | 165 | 65
  Conjunctival: No | 191 | 73 | 164 | 64
  Conjunctival: Yes | 0 | 3 | 1 | 1

36. Secondary Outcome: Total Number of Bleeding Events and Number of Each Type of Bleeding Events According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Total number of bleeding events and number of bleeding events for the following bleeding types is reported:
  * Intracranial
  * Digestive
  * Genitourinary
  * Gingival
  * Nasal
  * Pulmonary
  * Articular-muscular
  * Conjunctival.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
events
  Number of total bleeding events: number analyzed (Participants) | 191 | 76 | 166 | 65
  Number of total bleeding events | 0.10 (0.42) | 0.12 (0.36) | 0.48 (1.01) | 0.28 (0.82)
  Number of intracranial events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of intracranial events | 0.02 (0.12) | 0.03 (0.16) | 0.04 (0.20) | 0.02 (0.12)
  Number of digestive events: number analyzed (Participants) | 191 | 76 | 166 | 65
  Number of digestive events | 0.06 (0.36) | 0.04 (0.20) | 0.27 (0.80) | 0.06 (0.30)
  Number of genitourinary events: number analyzed (Participants) | 191 | 76 | 164 | 65
  Number of genitourinary events | 0.01 (0.10) | 0.00 (0.00) | 0.04 (0.19) | 0.06 (0.35)
  Number of gingival events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of gingival events | 0.00 (0.00) | 0.01 (0.11) | 0.01 (0.11) | 0.03 (0.25)
  Number of nasal events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of nasal events | 0.00 (0.00) | 0.00 (0.00) | 0.07 (0.36) | 0.08 (0.37)
  Number of pulmonary events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of pulmonary events | 0.00 (0.00) | 0.00 (0.00) | 0.02 (0.19) | 0.02 (0.12)
  Number of articular-muscular events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of articular-muscular events | 0.01 (0.10) | 0.00 (0.00) | 0.02 (0.19) | 0.00 (0.00)
  Number of conjunctival events: number analyzed (Participants) | 191 | 76 | 165 | 65
  Number of conjunctival events | 0.00 (0.00) | 0.04 (0.20) | 0.01 (0.08) | 0.02 (0.12)

37. Secondary Outcome: CHA2DS2-VASc Total Score According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category (CHA2DS2-VASc) score is a clinical prediction rule to estimate the risk of stroke in patients with Atrial Fibrillation (AF); it is frequently used to determine the need for an anticoagulation therapy, relating the high scores to a great risk of stroke and a low score corresponds to a lower risk of stroke. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
score on a scale | 4.05 (1.34) | 4.43 (1.33) | 4.63 (1.36) | 4.32 (1.28)

38. Secondary Outcome: Number of Patients on Each Category of CHA2DS2-VASc Score According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category (CHA2DS2-VASc) total score was categorized in three categories, according to the risk of stroke:
  * Low risk (score 0 in male; score 1 in female)
  * Moderate risk (score 1 in male; score 2 in female)
  * High risk (score ≥2 in male; score ≥3 in female)
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Low risk | 0 | 0 | 0 | 0
  Moderate risk | 0 | 0 | 0 | 0
  High risk | 192 | 76 | 166 | 66

39. Secondary Outcome: HAS-BLED Total Score According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile International Normalized Ratio (INR), Elderly (>65 years), Drugs and Alcohol (HAS-BLED) score may range from 0 to 9 with 0 being the best outcome. The high scores indicate a greater risk of bleeding and a low score corresponds to a lower risk of bleeding.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
score on a scale | 1.99 (0.82) | 1.64 (0.78) | 2.01 (0.92) | 2.06 (0.93)

40. Secondary Outcome: Number of Patients in Each Category of HAS-BLED Score According to Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: The Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol (HAS-BLED) total score was categorized in three categories according to the bleeding risk:
  * Low risk (score 0)
  * Intermediate risk (score 1-2)
  * High risk (score ≥3)
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Low risk | 0 | 0 | 0 | 0
  Intermediate risk | 147 | 64 | 118 | 48
  High risk | 45 | 12 | 48 | 18

41. Secondary Outcome: Number of Patients With Any Concomitant Treatments to Non-vitamin K Antagonist Oral Anticoagulant (NOAC) and Number of Patients for Each Concomitant Treatment to NOAC at Study Visit According to Current NOAC Type
Description: Number of patients in each category (No;Yes) of any concomitant treatments to NOAC and number of patients in each category (No; Yes) for each concomitant treatment to NOAC at study visit according to current NOAC type is reported.
  The concomitant treatment to non-vitamin K antagonist oral anticoagulant (NOAC) were the following:
  * Angiotensin-Receptor Blockers (ARB) or Angiotensin Converting Enzyme inhibitors (ACE) inhibitor
  * Beta-blocker
  * Calcium channel blockers
  * Diuretics
  * Amiodarone
  * Statin
  * Proton pump inhibitor
  * H2-receptor antagonist
  * Digoxin
  * NSAIDs (Nonsteroidal Anti-Inflammatory Drugs)
  * Dronedarone
  * Ketoconazole
  * Cyclosporine
  * Itraconazole
  * Other antiarrhythmics
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Any concomitant treatments to NOAC: No | 0 | 0 | 0 | 0
  Any concomitant treatments to NOAC: Yes | 192 | 76 | 166 | 66
  ARB or ACE inhibitor: No | 54 | 20 | 57 | 18
  ARB or ACE inhibitor: Yes | 138 | 56 | 109 | 48
  Beta-blocker: No | 82 | 27 | 54 | 21
  Beta-blocker: Yes | 110 | 49 | 112 | 45
  Calcium channel blockers: No | 154 | 53 | 136 | 47
  Calcium channel blockers: Yes | 38 | 23 | 30 | 19
  Diuretics: No | 87 | 32 | 56 | 19
  Diuretics: Yes | 105 | 44 | 110 | 47
  Amiodarone: No | 174 | 67 | 146 | 62
  Amiodarone: Yes | 18 | 9 | 20 | 4
  Statin: No | 83 | 34 | 77 | 18
  Statin: Yes | 109 | 42 | 89 | 48
  Proton pump inhibitor: No | 89 | 29 | 58 | 17
  Proton pump inhibitor: Yes | 103 | 47 | 108 | 49
  H2-receptor antagonist: No | 191 | 75 | 162 | 65
  H2-receptor antagonist: Yes | 1 | 1 | 4 | 1
  Digoxin: No | 168 | 71 | 153 | 57
  Digoxin: Yes | 24 | 5 | 13 | 9
  NSAIDs: No | 180 | 72 | 155 | 61
  NSAIDs: Yes | 12 | 4 | 11 | 5
  Dronedarone: No | 192 | 76 | 163 | 66
  Dronedarone: Yes | 0 | 0 | 3 | 0
  Ketoconazole: No | 192 | 76 | 166 | 66
  Ketoconazole: Yes | 0 | 0 | 0 | 0
  Cyclosporine: No | 192 | 76 | 166 | 66
  Cyclosporine: Yes | 0 | 0 | 0 | 0
  Itraconazole: No | 192 | 76 | 166 | 66
  Itraconazole: Yes | 0 | 0 | 0 | 0
  Other antiarrhythmics: No | 188 | 73 | 160 | 65
  Other antiarrhythmics: Yes | 4 | 3 | 6 | 1

42. Secondary Outcome: Number of Patients in Each Category of Previous Vitamin K Antagonists (VKA) Treatment According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Number of patients in each category of previous Vitamin K Antagonists (VKA) treatment according to duration since the first non-vitamin K antagonist oral anticoagulant (NOAC) initiation is reported.
  Previous VKA treatment was categorized in 2 categories:
  * No;
  * Yes.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- ≤4 Months: All patients who were on non-vitamin K antagonist oral anticoagulant (NOAC) ≤4 months.
- >4 Months: All patients who were on non-vitamin K antagonist oral anticoagulant (NOAC)>4 months.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  No | 26 | 187
  Yes | 13 | 274

43. Secondary Outcome: Number of Patients Treated Previously With the VKA Acenocoumarol and Number of Patients Treated Previously With the VKA Warfarin According to Duration Since the First NOAC Initiation
Description: Number of patients treated previously (before they were treated with non-vitamin K antagonist oral anticoagulant (NOAC)) with the Vitamin K Antagonists (VKA) acenocoumarol and number of patients treated previously with the VKA warfarin according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who previously received VKA treatment. One patient received acenocoumarol and warfarin during the study, so the total percentage is not 100%.
Measure: Count of Participants; unit: Participants
Groups:
- >4 Months: All patients who were on non-vitamin K antagonist oral anticoagulant (NOAC) >4 months.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 13 | 274
Participants
  Acenocoumarol | 13 | 263
  Warfarin | 0 | 12

44. Secondary Outcome: Duration of Previous Vitamin K Antagonists (VKA) Treatment According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Duration of treatment (in years) is reported for:
  * All patients treated previously with Vitamin K Antagonists (VKA) (row:All patients treated previously with VKA)
  * Patients treated only with the VKA warfarin (row: Warfarin patients)
  * Patients treated only with the VKA acenocoumarol (row: Acenocoumarol patients)
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 13 | 274
Years
  Acenocoumarol patients: number analyzed (Participants) | 12 | 259
  Acenocoumarol patients | 3.65 (3.85) | 3.88 (4.14)
  Warfarin patients: number analyzed (Participants) | 0 | 12
  Warfarin patients |  | 3.35 (1.94)
  All patients treated previously with VKA: number analyzed (Participants) | 12 | 270
  All patients treated previously with VKA | 3.65 (3.85) | 3.87 (4.07)

45. Secondary Outcome: Duration Since Non-valvular Atrial Fibrillation (NVAF) Diagnosis Until First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation According to Duration Since the First NOAC Initiation
Description: Duration (in years) since non-valvular atrial fibrillation (NVAF) diagnosis until first NOAC initiation according to duration since the first NOAC initiation is reported for:
  * All patients
  * Patients treated previously with VKA
  * Patients treated only with NOAC as anticoagulant (AC)
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 460
Years
  All patients | 1.62 (2.77) | 3.27 (4.95)
  Patients treated previously with VKA: number analyzed (Participants) | 13 | 273
  Patients treated previously with VKA | 3.71 (3.70) | 4.84 (4.79)
  Patients treated with NOAC as first AC: number analyzed (Participants) | 26 | 187
  Patients treated with NOAC as first AC | 0.58 (1.30) | 0.99 (4.27)

46. Secondary Outcome: First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Received and First NOAC Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who received dabigatran, rivaroxaban, apixaban, edoxaban as first NOAC and number of patients who received dabigatran 110 mg BID (twice daily), dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD as first NOAC according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  First NOAC received: Dabigatran ( 110 mg BID and 150 mg BID patients) | 23 | 174
  First NOAC received: Rivaroxaban (15 mg QD and 20 mg QD patients) | 2 | 81
  First NOAC received: Apixaban (2.5 mg BID and 5 mg BID patients) | 9 | 143
  First NOAC received: Edoxaban (30 mg QD and 60 mg QD patients) | 5 | 63
  First NOAC dose: Dabigatran 110 mg BID: number analyzed (Participants) | 23 | 174
  First NOAC dose: Dabigatran 110 mg BID | 6 | 88
  First NOAC dose: Dabigatran 150 mg BID: number analyzed (Participants) | 23 | 174
  First NOAC dose: Dabigatran 150 mg BID | 17 | 86
  First NOAC dose: Rivaroxaban 15 mg QD: number analyzed (Participants) | 2 | 81
  First NOAC dose: Rivaroxaban 15 mg QD | 0 | 30
  First NOAC dose: Rivaroxaban 20 mg QD: number analyzed (Participants) | 2 | 81
  First NOAC dose: Rivaroxaban 20 mg QD | 2 | 51
  First NOAC dose: Apixaban 2.5 mg BID: number analyzed (Participants) | 9 | 143
  First NOAC dose: Apixaban 2.5 mg BID | 4 | 53
  First NOAC dose: Apixaban 5 mg BID: number analyzed (Participants) | 9 | 143
  First NOAC dose: Apixaban 5 mg BID | 5 | 90
  First NOAC dose: Edoxaban 30 mg QD: number analyzed (Participants) | 5 | 63
  First NOAC dose: Edoxaban 30 mg QD | 4 | 26
  First NOAC dose: Edoxaban 60 mg QD: number analyzed (Participants) | 5 | 63
  First NOAC dose: Edoxaban 60 mg QD | 1 | 37

47. Secondary Outcome: Number of Patients Who Changed (Increased and Decreased) and Did Not Change the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who changed (increased and decreased) and did not change the first non-vitamin K antagonist oral anticoagulant (NOAC) dose according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- >4 Months: All patients who were on non-vitamin K antagonist oral anticoagulant (NOAC) ≤4 months.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  No | 39 | 427
  Yes (increase) | 0 | 8
  Yes (decrease) | 0 | 26

48. Secondary Outcome: First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Duration (in Years) According to Duration Since the First NOAC Initiation
Description: Treatment duration (in years) is reported for:
  * Patients who stopped first NOAC treatment;
  * Patients who did not stop the first NOAC treatment.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Years
  Patients who stopped first NOAC treatment: number analyzed (Participants) | 1 | 42
  Patients who stopped first NOAC treatment | 0.01 | 1.60 (1.61)
  Patients who did not stop the first NOAC treatment: number analyzed (Participants) | 38 | 419
  Patients who did not stop the first NOAC treatment | 0.30 (0.03) | 2.38 (1.93)

49. Secondary Outcome: Number of Patients in Each Category of Reason for First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Discontinuation According to Duration Since the First NOAC Initiation
Description: Reason for first NOAC treatment discontinuation was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Only patients who stopped first NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 1 | 42
Participants
  Lack of effectiveness | 0 | 1
  Investigator's decision | 0 | 15
  Patient's decision | 0 | 7
  Adverse event | 1 | 19

50. Secondary Outcome: Number of Patients in Each Category of Reason for First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Change Dose According to Duration Since the First NOAC Initiation
Description: Reason for first NOAC treatment change was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Only patients who changed dose in first NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 34
Participants
  Lack of effectiveness |  | 2
  Investigator's decision |  | 24
  Patient's decision |  | 0
  Adverse event |  | 8

51. Secondary Outcome: Number of Switches to a New Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Per Patient According to Duration Since the First NOAC Initiation
Description: Number of switches to a new non-vitamin K antagonist oral anticoagulant (NOAC) per patient according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: switches per patient
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
switches per patient | 0.03 (0.16) | 0.10 (0.35)

52. Secondary Outcome: Number of Patients in Each Category of Number of Switches to a New Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Per Patient According to Duration Since the First NOAC Initiation
Description: Number of patients based on the number of switches to a new NOAC per patient according to duration since the first NOAC initiation is reported.
  Number of switches to a new NOAC was categorized in 3 categories:
  * 0 switches
  * 1 switch
  * 2 switches.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  0 switches | 38 | 419
  1 switch | 1 | 36
  2 switches | 0 | 6

53. Secondary Outcome: Total Number of Switches According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Total number of switches according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who switched to a new NOAC.
Measure: Number; unit: Switches to a new NOAC
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 1 | 48
Switches to a new NOAC
  Dabigatran to Rivaroxaban | 0 | 3
  Dabigatran to Apixaban | 0 | 9
  Dabigatran to Edoxaban | 0 | 2
  Rivaroxaban to Dabigatran | 0 | 0
  Rivaroxaban to Apixaban | 1 | 10
  Rivaroxaban to Edoxaban | 0 | 2
  Apixaban to Dabigatran | 0 | 5
  Apixaban to Rivaroxaban | 0 | 3
  Apixaban to Edoxaban | 0 | 4
  Edoxaban to Dabigatran | 0 | 4
  Edoxaban to Rivaroxaban | 0 | 0
  Edoxaban to Apixaban | 0 | 6

54. Secondary Outcome: Number of Switches in Each Category of Reason for Switch According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Reason for switch was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who switched to a new NOAC.
Measure: Number; unit: Switches to another NOAC
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 1 | 48
Switches to another NOAC
  Lack of effectiveness | 0 | 1
  Investigator's decision | 0 | 17
  Patient's decision | 0 | 7
  Adverse event | 1 | 23

55. Secondary Outcome: Second Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Received and Second NOAC Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who received dabigatran, rivaroxaban, apixaban, edoxaban as second NOAC and number of patients who received dabigatran 110 mg BID (twice daily), dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD as second NOAC according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Number of patients who stopped the first NOAC treatment and switched to a second NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 1 | 42
Participants
  Second NOAC received: Dabigatran (110 mg BID and 150 mg BID patients) | 0 | 8
  Second NOAC received: Rivaroxaban (15 mg QD and 20 mg QD patients) | 0 | 5
  Second NOAC received: Apixaban (2.5 mg BID and 5 mg BID patients) | 1 | 21
  Second NOAC received: Edoxaban (30 mg QD and 60 mg QD patients) | 0 | 8
  Second NOAC dose: Dabigatran 110 mg BID: number analyzed (Participants) | 0 | 8
  Second NOAC dose: Dabigatran 110 mg BID |  | 6
  Second NOAC dose: Dabigatran 150 mg BID: number analyzed (Participants) | 0 | 8
  Second NOAC dose: Dabigatran 150 mg BID |  | 2
  Second NOAC dose: Rivaroxaban 15 mg QD: number analyzed (Participants) | 0 | 5
  Second NOAC dose: Rivaroxaban 15 mg QD |  | 3
  Second NOAC dose: Rivaroxaban 20 mg QD: number analyzed (Participants) | 0 | 5
  Second NOAC dose: Rivaroxaban 20 mg QD |  | 2
  Second NOAC dose: Apixaban 2.5 mg BID: number analyzed (Participants) | 1 | 21
  Second NOAC dose: Apixaban 2.5 mg BID | 0 | 13
  Second NOAC dose: Apixaban 5 mg BID: number analyzed (Participants) | 1 | 21
  Second NOAC dose: Apixaban 5 mg BID | 1 | 8
  Second NOAC dose: Edoxaban 30 mg QD: number analyzed (Participants) | 0 | 8
  Second NOAC dose: Edoxaban 30 mg QD |  | 3
  Second NOAC dose: Edoxaban 60 mg QD: number analyzed (Participants) | 0 | 8
  Second NOAC dose: Edoxaban 60 mg QD |  | 5

56. Secondary Outcome: Number of Patients Who Changed (Increased or Decreased) and Did Not Change the Second Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who changed (increased or decreased) and did not change the second non-vitamin K antagonist oral anticoagulant (NOAC) dose according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped the first NOAC treatment and switched to a second NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 1 | 42
Participants
  No | 1 | 40
  Yes (increase) | 0 | 1
  Yes (decrease) | 0 | 1

57. Secondary Outcome: Second Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Duration (in Years) According to Duration Since the First NOAC Initiation
Description: Second NOAC treatment duration (in years) according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped second NOAC treatment.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 6
Years |  | 0.49 (0.39)

58. Secondary Outcome: Number of Patients in Each Category of Reason for Second Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Discontinuation According to Duration Since the First NOAC Initiation
Description: Reason for second non-vitamin K antagonist oral anticoagulant (NOAC) treatment discontinuation was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped second NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 6
Participants
  Lack of effectiveness |  | 0
  Investigator's decision |  | 2
  Patient's decision |  | 0
  Adverse event |  | 4

59. Secondary Outcome: Number of Patients in Each Category of Reason for Second Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Change Dose According to Duration Since the First NOAC Initiation
Description: Reason for second NOAC treatment change was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who changed dose in second NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 2
Participants
  Lack of effectiveness |  | 0
  Investigator's decision |  | 2
  Patient's decision |  | 0
  Adverse event |  | 0

60. Secondary Outcome: Third Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Received and Third NOAC Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who received dabigatran, rivaroxaban, apixaban, edoxaban as third NOAC and number of patients who received dabigatran 110 mg BID (twice daily), dabigatran 150 mg BID, rivaroxaban 15 mg once daily (QD), rivaroxaban 20 mg QD, apixaban 2.5 mg BID, apixaban 5 mg BID, edoxaban 30 mg QD and edoxaban 60 mg QD as third NOAC according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped second NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 6
Participants
  Third NOAC received: Dabigatran |  | 1
  Third NOAC received: Rivaroxaban |  | 1
  Third NOAC received: Apixaban |  | 4
  Third NOAC received:Edoxaban |  | 0
  Third NOAC dose: Dabigatran 110 mg BID: number analyzed (Participants) | 0 | 1
  Third NOAC dose: Dabigatran 110 mg BID |  | 1
  Third NOAC dose: Dabigatran 150 mg BID: number analyzed (Participants) | 0 | 1
  Third NOAC dose: Dabigatran 150 mg BID |  | 0
  Third NOAC dose: Rivaroxaban 15 mg QD: number analyzed (Participants) | 0 | 1
  Third NOAC dose: Rivaroxaban 15 mg QD |  | 1
  Third NOAC dose: Rivaroxaban 20 mg QD: number analyzed (Participants) | 0 | 1
  Third NOAC dose: Rivaroxaban 20 mg QD |  | 0
  Third NOAC dose: Apixaban 2.5 mg BID: number analyzed (Participants) | 0 | 4
  Third NOAC dose: Apixaban 2.5 mg BID |  | 3
  Third NOAC dose: Apixaban 5 mg BID: number analyzed (Participants) | 0 | 4
  Third NOAC dose: Apixaban 5 mg BID |  | 1
  Third NOAC dose: Edoxaban 30 mg QD: number analyzed (Participants) | 0 | 0
  Third NOAC dose: Edoxaban 60 mg QD: number analyzed (Participants) | 0 | 0

61. Secondary Outcome: Number of Patients Who Changed (Increased and Decreased) and Did Not Change the Third Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Dose According to Duration Since the First NOAC Initiation
Description: Number of patients who changed (increased and decreased) and did not change the third non-vitamin K antagonist oral anticoagulant (NOAC) dose according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who started third NOAC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 6
Participants
  No |  | 6
  Yes (increase) |  | 0
  Yes (decrease) |  | 0

62. Secondary Outcome: Third Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Duration (in Years) According to Duration Since the First NOAC Initiation
Description: Duration of third NOAC treatment for patients who stopped NOAC treatment.
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped third NOAC treatment. No patient stopped the third NOAC treatment.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Number of Patients in Each Category of Reason for Third Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Discontinuation According to Duration Since the First NOAC Initiation
Description: Reason for Third NOAC treatment discontinuation was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who stopped third NOAC treatment. No patient stopped the third NOAC treatment.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Number of Patients in Each Category of Reason for Third Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment Change Dose According to Duration Since the First NOAC Initiation
Description: Reason for Third NOAC treatment change was categorized in four categories:
  * Lack of effectiveness
  * Investigator's decision
  * Patient's decision
  * Adverse event
Time Frame: At the single study visit (Day 1).
Population: Participants of FAS who changed dose in third NOAC treatment. No patients stopped the third NOAC treatment.
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Duration (in Years) in Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment According to Duration Since the First NOAC Initiation
Description: Duration (in years) in NOAC treatment is reported for:
  * All patients (patients who received or did not receive VKA)
  * Patients treated previously with Vitamin K Antagonists (VKA)
  * Patients treated with NOAC as first anticoagulant
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Years
  All patients | 0.29 (0.03) | 2.45 (1.96)
  Patients treated previously with VKA | 0.29 (0.03) | 2.39 (1.98)
  Patients treated with NOAC as first anticoagulant | 0.29 (0.03) | 2.54 (1.94)

66. Secondary Outcome: Number of Patients in Each Category of Total Time in Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Treatment According to Duration Since the First NOAC Initiation
Description: Number of patients in each category of total time in non-vitamin K antagonist oral anticoagulant (NOAC) treatment according to duration since the first NOAC initiation is reported.
  Total time in NOAC treatment was categorized in 4 categories:
  * <1 year;
  * 1-2 years;
  * 2-3 years;
  * >3 years.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  <1 year | 39 | 149
  1-2 years | 0 | 87
  2-3 years | 0 | 74
  >3 years | 0 | 151

67. Secondary Outcome: Number of Patients for Each Type of Antiplatelet Treatment According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Number of patients for each type of following antiplatelet treatment that the patients ever received is reported:
  * None (reports the patients who did not receive any antiplatelet treatment)
  * Acetyl salicylic acid
  * Clopidogrel
  * Prasugrel
  * Ticlopidine
  * Ticagrelor
  * Cilostazol
  * Triflusal
  * Dipyridamole
  * Others (other antiplatelet treatment than above mentioned).
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  None (no antiplatelet treatment received) | 35 | 314
  Acetyl salicylic acid | 4 | 124
  Clopidogrel | 1 | 43
  Prasugrel | 0 | 2
  Ticlopidine | 0 | 1
  Ticagrelor | 0 | 1
  Cilostazol | 0 | 0
  Triflusal | 0 | 3
  Dipyridamole | 0 | 0
  Others (other antiplatelet treatment than listed above) | 0 | 0

68. Secondary Outcome: Number of Patients for Each Type of Antiplatelet Treatment at the Time of Study Visit According to Duration Since the First NOAC Initiation
Description: Number of patients for each of the following antiplatelet treatment types at the time of study visit according to duration since the first NOAC initiation is reported:
  * None (reports the patients who did not receive any antiplatelet treatment)
  * Acetyl salicylic acid
  * Clopidogrel
  * Prasugrel
  * Ticlopidine
  * Ticagrelor
  * Cilostazol
  * Triflusal
  * Dipyridamole
  * Others (other antiplatelet treatment than above mentioned).
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Participants
  None | 38 | 444
  Acetyl salicylic acid | 0 | 9
  Clopidogrel | 1 | 11
  Prasugrel | 0 | 0
  Ticlopidine | 0 | 0
  Ticagrelor | 0 | 1
  Cilostazol | 0 | 0
  Triflusal | 0 | 3
  Dipyridamole | 0 | 0
  Others | 0 | 0

69. Secondary Outcome: Time in Treatment With Antiplatelet Agents (in Years) According to Duration Since the First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Initiation
Description: Time in treatment with antiplatelet agents (in years) according to duration since the first NOAC initiation is reported.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | ≤4 Months | >4 Months
Number analyzed (Participants) | 39 | 461
Years | 5.82 (1.66) | 5.98 (7.06)

70. Secondary Outcome: Number of Patients in Each Score of Clinical Frailty Scale Grading at the Time of the Study Visit According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Clinical Frailty Scale (CFS) is used commonly to assess frailty. It is a 9-point scale from 1 to 9 (1=very fit; 2=well; 3=Managing well; 4=Vulnerable; 5=Mildly frail; 6=Moderately frail; 7=Severely frail; 8=very severely frail; 9=terminally ill) that summarizes the overall level of fitness or frailty of an older adult after they had been evaluated by a health care professional. Applying the CFS to patients is quick and requires data collection by watching the patient (mobilize), inquiring about their habitual physical activity and ability. A person with a score >4 was considered frail.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  1-Very fit | 11 | 6 | 8 | 0
  2-Well | 24 | 15 | 18 | 9
  3-Managing well | 79 | 23 | 44 | 24
  4-Vulnerable | 45 | 11 | 46 | 19
  5-Mildly frail | 13 | 8 | 16 | 7
  6-Moderately frail | 15 | 10 | 24 | 3
  7-Severely frail | 4 | 3 | 9 | 3
  8-Very severely frail | 1 | 0 | 1 | 1
  9-Terminally ill | 0 | 0 | 0 | 0

71. Secondary Outcome: Number of Patients in Each Category Clinical Frailty Scale at the Time of the Study Visit According to Current Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Type
Description: Clinical Frailty Scale (CFS) is used commonly to assess frailty. It is a 9-point scale from 1 to 9 (1=very fit; 2=well; 3=Managing well; 4=Vulnerable; 5=Mildly frail; 6=Moderately frail; 7=Severely frail; 8=very severely frail; 9=terminally ill) that summarizes the overall level of fitness or frailty of an older adult after they had been evaluated by a health care professional. Applying the CFS to patients is quick and requires data collection by watching the patient (mobilize), inquiring about their habitual physical activity and ability.
  CFS was categorized in two categories, according to this ranges:
  * Frailty patients - CFS scoring >4
  * Non-frailty patients - CFS scoring ≤4
Time Frame: At the single study visit (Day 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 192 | 76 | 166 | 66
Participants
  Non-frailty patients (CFS scoring ≤4) | 159 | 55 | 116 | 52
  Frailty patients (CFS scoring >4) | 33 | 21 | 50 | 14

72. Secondary Outcome: Number of Patients in Each Category of Reason for First Non-vitamin K Antagonist Oral Anticoagulant (NOAC) Usage at the Time of First NOAC Initiation According to Current NOAC Type
Description: Reason for First NOAC usage was categorized in the following two categories:
  * Primary prevention;
  * Secondary prevention.
Time Frame: At the single study visit (Day 1).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Number analyzed (Participants) | 190 | 75 | 166 | 66
Participants
  Primary prevention | 138 | 61 | 135 | 54
  Secondary prevention | 52 | 14 | 31 | 12

ADVERSE EVENTS:
Time Frame: Information about the adverse events (AEs) was collected from the patients' medical records at the time of single study visit (Day 1). AEs collection covered a total time of 10 years.
Description: Adverse events were collected and reported only for patients who received dabigatran either as first NOAC, or second NOAC or third NOAC.For rivaroxaban, apixaban and edoxaban patients' adverse events were not assessed.
Groups:
- All Dabigatran Patients: This group included all patients who received dabigatran either as first NOAC (patients who the first NOAC prescribed was dabigatran), or as second NOAC (patients who stopped the first prescribed NOAC and received dabigatran as second NOAC), or as third NOAC (patients who stopped the second prescribed NOAC and received dabigatran as third NOAC).
Arm/Group | All Dabigatran Patients
All-Cause Mortality (participants affected / at risk) | 0/206
Serious Adverse Events (participants affected / at risk) | 4/206
Other Adverse Events (participants affected / at risk) | 0/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Dabigatran Patients (N=206)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT03993119/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03993119/SAP_001.pdf